CLINICAL TRIAL: NCT03967002
Title: Efficacy of Minimally Invasive Corticotomy Surgery in the Orthodontic Treatment of Mandibular Dental Crowding: A Randomized Prospective Study
Brief Title: Treatment of the Mandibular Dental Crowding With and Without Corticotomy Surgery
Acronym: CORTICO
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ardentis Cliniques Dentaires (Industry)
Collaborators: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Study CORTICO; 2019-00160 (Registry Identifier: CER-VD)
Record Dates: First submitted 2019-05-21; First posted 2019-05-29 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Dental Research; Orthodontics; Surgery, Oral; Maxillofacial Surgery; Tooth Disorder
Keywords: Accelerated orthodontics; Alveolar corticotomy; Piezoelectric surgery; Tooth movement; Dental crowding; Guided surgery; Minimally invasive oral surgery; Mandibular anterior alignment; Randomized prospective study
MeSH Terms: conditions — Tooth Diseases; Crowding

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test group with corticotomy surgery (Experimental): Orthodontic treatment and minimally invasive corticotomy surgery with piezoelectric device and surgical guide
  Interventions: Procedure: Test group with corticotomy surgery
- Control group without corticotomy surgery (No Intervention): Standard orthodontic treatment without surgery

INTERVENTIONS:
Procedure: Test group with corticotomy surgery — The surgery of corticotomy is performed with a piezo electric device and a personalized surgical guide just before the placement of orthodontic appliance. The initial impressions of the patient's dental arch as well as its three-dimensional radiography (CBCT) are used to create a perfectly adapted guide for minimally invasive corticotomy surgery.
  The incisions are made between the roots of:
  * the second premolars and first premolars,
  * the first lower premolars and canines,
  * the canines and lateral incisors,
  * the lateral incisors and central incisors, and,
  * the two lower central incisors.
  Arms: Test group with corticotomy surgery

SUMMARY:
The use of corticotomy surgery in addition to orthodontic standard treatment could accelerate the treatment. Corticotomy involves vertical interdental incisions of the gingiva and the bone with a very low thickness. Orthodontic appliances are placed immediately after the surgery.

This study aims to compare the tooth movement when correcting mandibular dental crowding in two groups of patients:

Test group: orthodontic treatment and minimally invasive corticotomy surgery. Control group: standard orthodontic treatment without surgery.

DETAILED DESCRIPTION:
Dental crowding in children, adolescents or adults is the most common reason to undergo orthodontic treatment. This malocclusion, characterized by the overlapping of teeth, is caused by a lack of space. In the mandibular anterior region, it is a predisposing factor for a periodontal disease. Good oral hygiene is difficult to maintain because the dental crowding promotes plaque retention in narrow interdental spaces and complicates the passage of brushes and dental floss. The standard orthodontic treatment lasts approximately 18-30 months. If the mandibular tooth space is less than 6 mm, it can be generally treated by orthodontics without therapeutic extractions.

Corticotomy has been a proven surgical technique for many years. It involves vertical interdental incisions of the gingiva and the bone with a very low thickness. It is mainly used to facilitate the movements of teeth. Dental movements associated with corticotomy may be twice as fast as those achieved with standard non-surgical treatment.

The study focuses on the correction of mandibular dental crowding. Its purpose is to compare the tooth movement obtained with orthodontic treatment and minimally invasive corticotomy surgery with that obtained with standard orthodontic treatment without surgery.

Patients requesting an orthodontic treatment to correct a dental crowding less than 12 mm are randomized to benefit from corticotomy surgery and orthodontic treatment (test group) or from only orthodontic treatment (control group). It is planned the inclusion of 22 patients, 11 in the test group and 11 in the control group.

After two visits necessary for the recruitment phase, treatment starts for the test group with the surgery and the appliance with brackets and arches, and, for the control group, with the appliance with brackets and arches.

The surgery of corticotomy is performed with a personalized surgical guide just before the placement of orthodontic appliance. The initial impressions of the patient's dental arch as well as its three-dimensional radiography (CBCT) make it possible to create a perfectly adapted guide. The incisions are made with a piezoelectric device between the roots of teeth, from the mandibular second premolar to the contralateral second mandibular premolar.

The study lasts 12 months after the placement of orthodontic material. During this 12 months, periodical controls (1 week, 2 weeks and 1-12 months) are carried out. After these 12 months, all patients undergo treatment with controls specific to standard orthodontic procedure.

ELIGIBILITY:
Inclusion Criteria:

* The patient is over 18 years old,
* The dental crowding of the patient does not exceed 12 mm. The crowding, measured from the right mandibular canine to the left mandibular canine, doesn't require extraction or orthognathic surgery.
* The patient has no active periodontal disease and no history of treated periodontal disease.
* The patient has good dental hygiene.
* The patient has no untreated decay.
* The patient accepts the wear of metallic orthodontic materials.

Exclusion Criteria:

The patient :

* is not able to understand the information given by the practitioner for legal, psychological or linguistic reasons.
* will have predictable follow-up difficulties.
* is pregnant.
* has a high risk of endocarditis.
* has severe or acquired immune deficiency.
* has a malignant condition, an history of radiotherapy in the mandibular region.
* has severe hematology, hemophilia, chronic renal failure, autoimmune disease, a condition requiring organ transplantation, poorly controlled diabetes, osteoporosis, rheumatoid arthritis or psychiatric illness.
* is under antimitotic, immunosuppressive or high dose corticosteroid treatment.
* smokes more than 10 cigarettes per day.
* has a systemic disease that affects bone, such as osteoporosis, hyperparathyroidism, or vitamin D deficiency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline tooth alignment at 12 months during the correction of the crowding in the anterior mandible. | Baseline, 2 weeks, and 1, 2, 3, 4, 5, 6 and 12 months
  The linear displacement (canine-to-canine) in millimeter of the anatomic contact points of each incisor from the anatomic point of the adjacent teeth is measured (method of irregularity index scoring of Little) on dental impressions with an electronic calipers.
  Total alignment between 0 (total alignment) and 6 (no alignment).

SECONDARY OUTCOMES:
Change from baseline plaque index at 12 months. | Baseline, 6 and 12 months
  The plaque index is scored using a periodontal probe at four sites around each tooth (mesial, distal, vestibular, palatal sides) and the average value is calculated. The range of the score is 0 to 3:
  score 0: No plaque; score 1: Plaque revealed with the use of probe on the tooth surface. Thin film of plaque.
  score 2: Plaque observed with naked eye. Moderate accumulation of soft deposit. score 3: Abundance of soft matter. Large amount of plaque.
Change from baseline modified sulcus bleeding index at 12 months. | Baseline, 6 and 12 months
  The modified sulcus bleeding index is scored using a periodontal probe at four sites around each tooth (mesial, distal, vestibular, palatal sides) and the average value is calculated. The range of the score is 0 to 3:
  score 0: No bleeding when a periodontal probe is passed along the gingival margin adjacent to the tooth; score 1: Isolated bleeding; score 2: Blood forms a confluent red line on margin; score 3: Heavy or profuse bleeding.
Change from baseline pocket probing depth at 12 months. | Baseline, 6 and 12 months
  The pocket probing depth measurement in millimeter is performed from the gingival margin to the epithelial attachment using a periodontal probe at four sites around each tooth (mesial, distal, vestibular, palatal sides) and the average value is calculated.
  It was classified as: no/mild pocket depth ≤3 mm, moderate pocket depth 4-5 mm, severe pocket depth ≥6 mm.
Change from baseline bone levels to 6 months. | Baseline and 6 months
  Measurement of height and thickness of the alveolar bone in millimeter using cone-beam computerized tomography (CBCT).
Time-to-event of complications and adverse events | Baseline, after surgery, after appliance of orthodontic material, 1 week, 2 weeks, and 1, 2, 3, 4, 5, 6 and 12 months
  The number and nature of complications and adverse events will be recorded at each visit and compared between interventional and control groups.
Pain intensity measures: analog visual scale | Baseline, after surgery, after appliance of orthodontic material, 1 week, 2 weeks, and 1, 2, 3, 4, 5, 6 and 12 months
  Self reported pain intensity at each visit. It is scored 0-10 with an analog visual scale. The score is determined by measuring the distance in centimeter on the 10-cm line between the "no pain" anchor (score 0) and the patient's mark, providing a range of scores from 0-10. The maximum of pain is scored 10.
  The mean of pain intensities of all patients at each control will be classified according to the following cut points:
  0-0.4 cm: no pain, 0.5-4.4 cm: mild pain, 4.5-7.4 cm: moderate pain, and 7.5-10 cm: severe pain.
Satisfaction measures: analog visual scale | 6 and 12 months
  Self reported satisfaction towards the treatment at the end of the treatment. It is scored 0-10 with an analog visual scale. The score is determined by measuring the distance in centimeter on the 10-cm line between the "no satisfaction" anchor (score 0) and the patient's mark, providing a range of scores from 0-10. The maximum of satisfaction is scored 10.
  The mean of satisfaction intensities of all patients at each control will be classified according to the following cut points:
  0-0.4 cm: no satisfaction, 0.5-4.4 cm: low satisfaction, 4.5-7.4 cm: moderate satisfaction, and 7.5-10 cm: high satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Marion Paris, DMD, Principal Investigator — Oral surgeon
Locations (1):
- Ardentis Clinique Dentaire, Écublens, Switzerland